CLINICAL TRIAL: NCT00720967
Title: Influence of Preoperative Hemodialysis or Intraoperative Modified Ultrafiltration on Postoperative Outcome for Patients With Severe Renal Dysfunction Undergoing Open Heart Surgery: Randomized, Controlled, Multicenter Clinical Trial
Brief Title: Preop Hemodialysis or Intraop Ultrafiltration for Patients With Severe Renal Dysfunction Undergoing Open Heart Surgery
Acronym: SeRenaD-CPB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Gaziantep (Other); Ankara University (Other); Pamukkale University (Other); German Heart Institute (Other); Hospices Civils de Lyon (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Erman Pektok, MD, University Hospital of Geneva, Service for Cardiovascular Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-058 (NAC 08018)
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2008-07-23 (Estimated); Status verified 2008-07

CONDITIONS: Non-Dialysis Dependent Severe Renal Dysfunction; Cardiovascular Disease
Keywords: Renal dysfunction; Hemodialysis; Modified ultrafiltration; Open heart surgery
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Control Group (Open heart surgery alone)
  Interventions: Procedure: Open Heart Surgery (OHS)
- 2 (Experimental): Intraoperative Modified Ultrafiltration (MUF) Group (Open heart surgery with intraoperative MUF)
  Interventions: Procedure: Open Heart Surgery (OHS); Procedure: Intraoperative Modified Ultrafiltration (MUF)
- 3 (Experimental): Preoperative Hemodialysis Group (Open Heart Surgery after preoperative hemodialysis)
  Interventions: Procedure: Open Heart Surgery (OHS); Procedure: Hemodialysis (HD)

INTERVENTIONS:
Procedure: Open Heart Surgery (OHS) — General anesthesia, use of iodine impregnated adhesive dressing, median sternotomy and/or thoracotomy incision, full heparinization (300-400 ui/kg), arterial and venous cannulation, initialization of CPB with or without aortic cross-clamping and high-potassium cold cardioplegia, surgical repair under mild-moderate hypothermia. De-clamping (if cross clamp was applied), neutralization of heparin by protamin, de-cannulation and hemostasis after surgical repair. Insertion of drain(s) and pacing wire(s). Closure of all layers in anatomical plan.
Procedure: Intraoperative Modified Ultrafiltration (MUF) — Once the surgical repair is finished, and CPB will be stopped after aortic declamping. The arterial and venous cannulae will be connected to each other using 3-way connectors and a cardioplegia line. When hemodynamic stability is established (MAP >75 mmHg, CVP > 12 mmHg, Htc > 25%), blood will be drained from the arterial cannula using a roller pump, driven to the ultrafilter, and eventually to the venous cannula. The blood flow will be maintained at ~150 mL/min, and suction will be applied to the filtrate port to achieve an ultrafiltration of 100-120 mL/min. Heat exchanger and bubble trap of the cardioplegia line will be used to maintain the filtered blood at body temperature and to prevent air embolism, respectively. MUF will continue 20 minutes. The filtered volume will be collected.
  Arms: 2
Procedure: Hemodialysis (HD) — Two HD sessions will be performed at 3 days and 1 day prior to surgery. Each session will last 3 hours if the patient weighs < 75 kg, and 4 hours if > 75 kg. Conventional HD will be carried out using a volume-controlled dialysis machine. A bicarbonate dialysate containing K (3 mmol/L), Ca (1.5 mmol/L) and HCO3 (31 mmol/L) will be used. Sodium conductivity will be set at 138 mmol/L. Medium-flow filters will be used as artificial kidney devices. Dialysate temperature will be set at 36oC. Dialysate and blood flow rate will be set at 500 mL/min and 250-300 ml/min, respectively. Intradialytic ultrafiltration will not be used routinely unless the patient has volume overload. The decision to use intradialytic ultrafiltration will be taken with the anaesthesiologist and the cardiac surgeon. If intradialytic ultrafiltration is indicated, maximal rate of ultrafiltration will be 10 ml/kg/hour. These patients will undergo open heart surgery after two sessions of HD.
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether preoperative hemodialysis or intraoperative modified ultrafiltration are effective for patients with non-dialysis dependent severe renal dysfunction undergoing open heart surgery.

DETAILED DESCRIPTION:
1. BACKGROUND

1.1. RENAL DYSFUNCTION AND OPEN HEART SURGERY:

The incidences of both cardiovascular disease (CVD) and chronic renal dysfunction (RD) are increasing with the aging population in the western world (1). The intense relationship between the pathogenesis of CVD and chronic RD has recently been reviewed by Schiffrin et al, in detail (2). They both have common risk factors such as diabetes, hypertension, activation of renin-angiotensin system, endothelial dysfunction, oxydative stress, etc. Besides, each has an impact on the other's outcome. On the one hand, CVD is the most frequent cause of death in chronic RD patients (3). On the other hand, even mild chronic RD is one of the major risk factors of postoperative mortality and morbidity after cardiac operations (4, 5). The mechanism is not clear yet, however, volume overload, electrolyte imbalance and inflammatory state created by cardiopulmonary bypass (CPB) may have an impact. Zakeri et al showed that in-hospital mortality after isolated primary coronary artery bypass grafting (CABG) increases exponentially with increasing levels of renal dysfunction (6). They reported an in-hospital mortality of 2.2%, 4.3%, 9.3% and 14.8% in patients who have a preoperative serum creatinine level (SCr) of <130 µmol/L, 130-149 µmol/L, 150-179 µmol/L and 180-199 µmol/L, respectively. These results were similar to the study published previously by Weerasinghe et al with the same cut-off levels of SCr (7). Using the Glomerular Filtration Rate (GFR) instead of SCr, Cooper et al. came to the same conclusion after analysing 483,914 patients receiving isolated CABG in the Society of Thoracic Surgeons (STS) National Adult Cardiac Database (5). They reported that operative mortality rose inversely with declining renal function, from 1.3% for those with normal renal function to 1.8%, 4.3% and 9.3% for patients with mild, moderate and severe RD, respectively. Another study regarding the effect of preoperative RD on mortality after valve surgery was also published with a relatively smaller patient population (8). Although the RD group had significantly worse outcomes with regard to postoperative ventilation time, re-operation, blood transfusion and length of hospital stay, operative mortality was not statistically different between the two groups (3.4% for RD group vs. 2.3% for the control group), probably because of small sample size. However, Filsoufi et al. reported an increased mortality for patients having SCr of >2.5 mg/dL after single valve replacement (25.0% vs. 2.4%),multiple valve replacement (26.7% vs. 3.4%), and combined valve replacement with CABG (28.0% vs. 4.6%) in a large, single-center cohort (9). Regarding long-term survival, Devbhandari reported 1-, 3- and 5-year survival rates following on-pump coronary bypass surgery as 90.3%, 83.2% and 71.4% for non-dialysis dependent renal dysfunction (NDDRD) patients, and 97.4%, 94.6% and 91.0% for patients with no history of RD, respectively (10). Chronic RD affects not only the operative mortality, but also the morbidity after open heart surgery. It has been shown that preoperative RD is an independent predictor of postoperative acute RD and hemodialysis (HD) (5, 7, 9-12) as well as gastrointestinal (GI) (4, 9), respiratory (5, 9), infectious (5) and neurological (5) complications.

1.2. HEMODIALYSIS:

HD is the most common renal replacement therapy for decades, for those who have end-stage RD and have not received renal transplantation. Intermittent HD is a very efficient method to decrease blood urea and creatinine as well as to treat volume overload. Intermittent HD can be performed temporarily in the setting of acute RD or permanently in the setting of chronic RD. In chronic RD, 3 sessions of 4 hours are usually prescribed to adequately substitute the renal function. A good vascular access is essential to perform HD. A temporary dual- or tri-lumen dialysis catheter has to be inserted into a central vein such as the internal jugular, the subclavian or the femoral vein.

1.3. ULTRAFILTRATION:

Intraoperative ultrafiltration has been used widely in pediatric open heart surgery for decades, reducing total body water, increasing hematocrit (Htc) levels, removing inflammatory mediators, thus improving the operative outcome (13). In the 90's, Naik et al. modified the technique (14), and reported better outcomes with modified ultrafiltration (MUF) in pediatric population (15). However, use of MUF has been limited to end-stage RD patients with volume overload undergoing open heart surgery, as an adjunct to pre- and postoperative HD in the adult population. The Verona group reported fewer respiratory, neurological, GI complications, and less blood product transfusion in the group of patients who received MUF after CPB, however mortality, overall morbidity, length of Intensive Care Unit (ICU) stay and length of hospital stay were comparable between MUF and control groups including 573 consecutive patients (16). A meta-analysis evaluating the effects of ultrafiltration on postoperative blood product use and perioperative bleeding in adult patients revealed fewer bleeding complications and reduced blood product use after intraoperative ultrafiltration (17). Boga et al reported improved cardiac performance after CABG surgery with MUF. However, they could not find any difference in Interleukin-6, Interleukin-8 and Neopterin levels. They attributed this effect to prevention of hemodilution and hypervolemia (18). In summary, no clear evidence is available at the present regarding the impact of intraoperative MUF on the operative outcome of NDDRD patients undergoing open heart surgery. Capuano et al. recently (19) reported successful results in a NDDRD patient who required urgent coronary revascularisation. Nevertheless, the impact of intraoperative MUF on the outcome of NDDRD patients undergoing open heart surgery remains unclear, and is worth investigation.

1.4. PREVIOUS STUDIES:

The quest to improve the outcome of NDDRD patients undergoing open heart surgery has been in the agenda of some groups to date. Two pioneering studies were recently published from Turkey (20, 21). The target patient population was NDDRD patients undergoing elective isolated primary CABG surgery. Patients were randomized into two groups prospectively, one group received 2 doses of prophylactic HD just before surgery whereas the other did not, and served as control. Both studies reported reduced operative mortality rates, reduced postoperative need for HD, and shorter length of stay in the prophylactic HD groups. However, these two studies had very limited number of patients with a short period of follow-up, excluded valve surgery, and did not analyse cost-effectiveness. Furthermore, intraoperative ultrafiltration was not studied.

1.5. ASSESSMENT OF RENAL FUNCTION:

GFR is the best measure of overall kidney function (22). The Cockroft-Gault formula is a commonly used way to predict GFR (23). GFR <30 mL/min/1.73 m2 is accepted as "severe RD" (22). SCr is a simple and practical universal biologic marker used for estimating glomerular filtration. Although SCr does not have a linear association with GFR, it has also been reported to be a powerful predictor of operative mortality (6). Thus, SCr and GFR were both accepted as preoperative indicators of RD with the cut-off levels of 180 µmol/L (or 2.0 mg/dL) and 30 mL/min/1.73 m2, respectively.

1.6. CONCLUSION:

In summary, this data mandates us a well defined strategy for patients with NDDRD in order to obtain better operative outcome. Under the guidance of the current literature, a randomized controlled trial (RCT) with a larger number of patients undergoing open heart surgery will provide precise answers for these questions. Comparison of hospital costs may add an extra value for the assessment of cost-effectiveness as well.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of SCr > 180 µmol/L or 2.0 mg/dL, and/or a GFR < 30 mL/min/1.73 m2.
* Indication for elective open heart surgery under CPB.

Exclusion Criteria:

* History of chronic or recent HD.
* Emergency status.
* Off-pump surgery.
* Failure to obtain patient consent documented by a signed consent form.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Operative mortality, defined as any death occurring within 30 days after the operation or any death occurring before discharge during the same hospitalization (in percentage). | within the first 30 days after surgery or before the discharge after surgery

SECONDARY OUTCOMES:
Survival at one year after surgery (in percentage). | one year after surgery
Postoperative low cardiac output (in percentage). | within the first 30 days after surgery or before the discharge after surgery
Postoperative permanent neurological deficit (in percentage). | within the first 30 days after surgery or before the discharge after surgery
Postoperative transient neurological deficit (in percentage). | within the first 30 days after surgery or before the discharge after surgery
Postoperative acute renal dysfunction (in percentage). | within the first 30 days after surgery or before the discharge after surgery
Postoperative persistent renal dysfunction requiring hemodialysis (in percentage). | within the first 30 days after surgery or before the discharge after surgery
Postoperative gastrointestinal complication (in percentage). | within the first 30 days after surgery or before the discharge after surgery
Postoperative respiratory failure (in percentage). | within the first 30 days after surgery or before the discharge after surgery
Postoperative systemic infection (in percentage). | within the first 30 days after surgery or before the discharge after surgery
Postoperative local infection (in percentage). | within the first 30 days after surgery or before the discharge after surgery
Postoperative new-onset arrythmia (in percentage). | within the first 30 days after surgery or before the discharge after surgery
Postoperative surgical drainage (in mL). | within the first 72 hours after surgery
Postoperative need for transfusion of blood products (in unit packs). | within the first 72 hours after surgery
Postoperative length of ICU stay (in days) | within the first 30 days after surgery or before the discharge after surgery
Postoperative length of hospital stay (in days) | within the first 30 days after surgery or before the discharge after surgery
Total hospital costs for the admission of operation (in Euros) | From the day of admission to hospital until the day of discharge after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Erman Pektok, MD, Principal Investigator — University Hospital of Geneva, Service for Cardiovascular Surgery; Patrick O Myers, MD, Study Director — University Hospital of Geneva, Service for Cardiovascular Surgery; Thomas Perneger, MD, PhD, Study Director — University Hospital of Geneva, Center of Clinical Research; Afksendiyos Kalangos, MD, PhD, Study Chair — University Hospital of Geneva, Service for Cardiovascular Surgery
Locations (7):
- University of Lyon, Hopital Cardiothoracique Louis Pradel, Lyon, France
- German Heart Institute Berlin, Berlin, Germany
- Hospital Clinico, University of Barcelona, Department of Cardiovascular Surgery, Barcelona, Spain
- University Hospital of Geneva, Service for Cardiovascular Surgery, Geneva, Switzerland
- Turkey (Türkiye) (3):
  - Ankara University, Department of Cardiovascular Surgery, Ankara
  - Pamukkale University, Department of Cardiovascular Surgery, Denizli
  - Gaziantep University, Department of Cardiovascular Surgery, Gaziantep

REFERENCES:
- [Background] Foley RN, Parfrey PS, Sarnak MJ. Epidemiology of cardiovascular disease in chronic renal disease. J Am Soc Nephrol. 1998 Dec;9(12 Suppl):S16-23. PMID 11443763
- [Background] Schiffrin EL, Lipman ML, Mann JF. Chronic kidney disease: effects on the cardiovascular system. Circulation. 2007 Jul 3;116(1):85-97. doi: 10.1161/CIRCULATIONAHA.106.678342. PMID 17606856
- [Background] Levin A, Foley RN. Cardiovascular disease in chronic renal insufficiency. Am J Kidney Dis. 2000 Dec;36(6 Suppl 3):S24-30. doi: 10.1053/ajkd.2000.19928. PMID 11118155
- [Background] Anderson RJ, O'brien M, MaWhinney S, VillaNueva CB, Moritz TE, Sethi GK, Henderson WG, Hammermeister KE, Grover FL, Shroyer AL. Renal failure predisposes patients to adverse outcome after coronary artery bypass surgery. VA Cooperative Study #5. Kidney Int. 1999 Mar;55(3):1057-62. doi: 10.1046/j.1523-1755.1999.0550031057.x. PMID 10027944
- [Background] Cooper WA, O'Brien SM, Thourani VH, Guyton RA, Bridges CR, Szczech LA, Petersen R, Peterson ED. Impact of renal dysfunction on outcomes of coronary artery bypass surgery: results from the Society of Thoracic Surgeons National Adult Cardiac Database. Circulation. 2006 Feb 28;113(8):1063-70. doi: 10.1161/CIRCULATIONAHA.105.580084. Epub 2006 Feb 20. PMID 16490821
- [Background] Zakeri R, Freemantle N, Barnett V, Lipkin GW, Bonser RS, Graham TR, Rooney SJ, Wilson IC, Cramb R, Keogh BE, Pagano D. Relation between mild renal dysfunction and outcomes after coronary artery bypass grafting. Circulation. 2005 Aug 30;112(9 Suppl):I270-5. doi: 10.1161/CIRCULATIONAHA.104.522623. PMID 16159830
- [Background] Weerasinghe A, Hornick P, Smith P, Taylor K, Ratnatunga C. Coronary artery bypass grafting in non-dialysis-dependent mild-to-moderate renal dysfunction. J Thorac Cardiovasc Surg. 2001 Jun;121(6):1083-9. doi: 10.1067/mtc.2001.113022. PMID 11385375
- [Background] Ibanez J, Riera M, Saez de Ibarra JI, Carrillo A, Fernandez R, Herrero J, Fiol M, Bonnin O. Effect of preoperative mild renal dysfunction on mortality and morbidity following valve cardiac surgery. Interact Cardiovasc Thorac Surg. 2007 Dec;6(6):748-52. doi: 10.1510/icvts.2007.159392. Epub 2007 Sep 21. PMID 17890235
- [Background] Filsoufi F, Rahmanian PB, Castillo JG, Chikwe J, Carpentier A, Adams DH. Early and late outcomes of cardiac surgery in patients with moderate to severe preoperative renal dysfunction without dialysis. Interact Cardiovasc Thorac Surg. 2008 Feb;7(1):90-5. doi: 10.1510/icvts.2007.164483. Epub 2007 Nov 22. PMID 18033787
- [Background] Devbhandari MP, Duncan AJ, Grayson AD, Fabri BM, Keenan DJ, Bridgewater B, Jones MT, Au J; North West Quality Improvement Programme in Cardiac Interventions. Effect of risk-adjusted, non-dialysis-dependent renal dysfunction on mortality and morbidity following coronary artery bypass surgery: a multi-centre study. Eur J Cardiothorac Surg. 2006 Jun;29(6):964-70. doi: 10.1016/j.ejcts.2006.03.038. Epub 2006 May 3. PMID 16675230
- [Background] Kilo J, Margreiter JE, Ruttmann E, Laufer G, Bonatti JO. Slightly elevated serum creatinine predicts renal failure requiring hemofiltration after cardiac surgery. Heart Surg Forum. 2005;8(1):E34-8. doi: 10.1532/HSF98.20041117. PMID 15769711
- [Background] Mangano CM, Diamondstone LS, Ramsay JG, Aggarwal A, Herskowitz A, Mangano DT. Renal dysfunction after myocardial revascularization: risk factors, adverse outcomes, and hospital resource utilization. The Multicenter Study of Perioperative Ischemia Research Group. Ann Intern Med. 1998 Feb 1;128(3):194-203. doi: 10.7326/0003-4819-128-3-199802010-00005. PMID 9454527
- [Background] Shen I, Giacomuzzi C, Ungerleider RM. Current strategies for optimizing the use of cardiopulmonary bypass in neonates and infants. Ann Thorac Surg. 2003 Feb;75(2):S729-34. doi: 10.1016/s0003-4975(02)04697-0. PMID 12607719
- [Background] Naik SK, Knight A, Elliott MJ. A successful modification of ultrafiltration for cardiopulmonary bypass in children. Perfusion. 1991;6(1):41-50. doi: 10.1177/026765919100600106. PMID 10149499
- [Background] Naik SK, Knight A, Elliott M. A prospective randomized study of a modified technique of ultrafiltration during pediatric open-heart surgery. Circulation. 1991 Nov;84(5 Suppl):III422-31. PMID 1934440
- [Background] Luciani GB, Menon T, Vecchi B, Auriemma S, Mazzucco A. Modified ultrafiltration reduces morbidity after adult cardiac operations: a prospective, randomized clinical trial. Circulation. 2001 Sep 18;104(12 Suppl 1):I253-9. doi: 10.1161/hc37t1.094931. PMID 11568065
- [Background] Boodhwani M, Williams K, Babaev A, Gill G, Saleem N, Rubens FD. Ultrafiltration reduces blood transfusions following cardiac surgery: A meta-analysis. Eur J Cardiothorac Surg. 2006 Dec;30(6):892-7. doi: 10.1016/j.ejcts.2006.09.014. Epub 2006 Oct 13. PMID 17046273
- [Background] Boga M, Islamoglu, Badak I, Cikirikcioglu M, Bakalim T, Yagdi T, Buket S, Hamulu A. The effects of modified hemofiltration on inflammatory mediators and cardiac performance in coronary artery bypass grafting. Perfusion. 2000 Mar;15(2):143-50. doi: 10.1177/026765910001500209. PMID 10789569
- [Background] Capuano F, Bianchini R, Goracci M, Roscitano A, Luciani R, Simon C, Giusti L, Sinatra R. Intraoperative veno-arterial hemofiltration during miniaturized extracorporeal bypass. Ann Thorac Surg. 2007 Jun;83(6):2215-6. doi: 10.1016/j.athoracsur.2006.12.002. PMID 17532433
- [Background] Durmaz I, Yagdi T, Calkavur T, Mahmudov R, Apaydin AZ, Posacioglu H, Atay Y, Engin C. Prophylactic dialysis in patients with renal dysfunction undergoing on-pump coronary artery bypass surgery. Ann Thorac Surg. 2003 Mar;75(3):859-64. doi: 10.1016/s0003-4975(02)04635-0. PMID 12645707
- [Background] Bingol H, Akay HT, Iyem H, Bolcal C, Oz K, Sirin G, Demirkilic U, Tatar H. Prophylactic dialysis in elderly patients undergoing coronary bypass surgery. Ther Apher Dial. 2007 Feb;11(1):30-5. doi: 10.1111/j.1744-9987.2007.00452.x. PMID 17309572
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066